CLINICAL TRIAL: NCT06267820
Title: A Comparative Study Between Combined Ketorolac Bupivacaine and Bupivacaine Alone for Transversus Abdominis Plane Block in Children Undergoing Lower Abdominal Surgeries: A Prospective Double- Blind Randomized Clinical Trial
Brief Title: Combined Ketorolac Bupivacaine Versus Bupivacaine Alone for TAP Block in Children Undergoing Lower Abdominal Surgeries
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Fouad Soliman, Lecturer of Anesthesia and ICU, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 2010
Record Dates: First submitted 2023-12-13; First posted 2024-02-20 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Postoperative Pain, Acute
Keywords: TAP; ketorolac; bupivacaine,; ultrasound; children
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Ketorolac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP block with bupivacaine and ketorolac (Active Comparator): Ultrasound guided TAP block with bupivacaine 0.25% (0.5 ml/kg) and ketorolac (0.5 mg/kg).
  Interventions: Drug: Bupivacain; Drug: Ketorolac
- TAP block with bupivacaine (Active Comparator): ultrasound guided TAP block with bupivacaine 0.25% (0.5 ml/kg).
  Interventions: Drug: Bupivacain

INTERVENTIONS:
Drug: Bupivacain — analgesia
  Other Names: bupivacaine
Drug: Ketorolac — analgesia
  Arms: TAP block with bupivacaine and ketorolac

SUMMARY:
Control of of pain in children is fundamental. TAP block is associated with less side effects compared with other neuraxial techniques especially when done under ultrasound guidance.

Ketorolac has analgesic effect comparable to morphine. Children were arranged randomly into two equal groups, forty-five children in each.

Group (K) (n= 45): received ultrasound guided TAP block with bupivacaine 0.25% (0.5 ml/kg) and ketorolac (0.5 mg/kg).

Group (T) (n =45): received ultrasound guided TAP block with bupivacaine 0.25% (0.5 ml/kg)

DETAILED DESCRIPTION:
This prospective randomized controlled study were carried out in Sohag university hospitals after getting approval from medical research ethics committee and written informed consents from the patients' parents or legal guardians. This study included 90 ASA status I and II children aged 6-12 years undergoing elective lower abdominal surgeries.Preoperative assessment:

* History taking from the parents.
* Complete physical examination.
* Laboratory investigations: Complete Blood Picture and coagulation profile. Preoperative preparation

Before starting, standard monitoring will be as follow:

1. Non-invasive blood pressure (systolic and diastolic).
2. Peripheral Oxygen saturation (SpO2%). After insertion of intravenous line, all children will receive atropine premedication (0.01-0.02 mg/kg). General anesthesia will be induced using propofol 1% (2 mg/kg), atracurium (0.5 mg/kg) to facilitate endotracheal intubation. Anesthesia will be maintained using isoflurane (1-2%) with controlled ventilation.At the end of operation, muscle relaxant is reversed using neostigmine and atropine.

Intraoperative hemodynamic parameters will be recorded throughout the surgery at fixed intervals (at time of skin incision then after every 5 min till the end of surgery).

Then TAP block were done under ultrasound guidance using either bupivacaine and ketorolac or bupivacaine alone

ELIGIBILITY:
Inclusion Criteria:

* ASA status I and II children Age 6-12 years Elective lower abdominal surgeries.

Exclusion Criteria:

* Parents' or legal guardians' refusal.
* A history of developmental delay or mental retardation.
* ASA III and IV.
* A known allergy to ketorolac or bupivacaine.
* Hemodynamic unstable patient
* Urgent surgeries

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
1st analgesic requirement | 24 hours
  the time at which the 1st need for analgesia is given.
Number of patients who requested analgesia | 24 hours
  Number (percentage)of patients who requested analgesia

SECONDARY OUTCOMES:
heart rate | 24 hours
  the patient vital sign (beats/min)
Total rescue analgesia | 24 hours
  Total rescue analgesia in the first 24 h. postoperatively
Satisfaction of the parents regarding their children analgesia | 24 hours
  using 5- point satisfaction scale (1= Very satisfied, 2=Satisfied,3= Neither satisfied nor dissatisfied,4= Dissatisfied, 5= Very dissatisfied).
  This satisfaction will be done by parents according to the VAS, incidence of side effects and analgesic requirements
Number of children in each group who required analgesia in the first 24 h postoperatively | 24 hours
  Number of children in each group who required analgesia in the first 24h postoperatively
blood pressure | 24 hours
  The patients blood pressure (mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Fouad I Soliman, MD, Principal Investigator — Sohag University
Locations (1):
- Fouad Ibrahim Soliman, Sohag, Egypt